CLINICAL TRIAL: NCT07242885
Title: The Effect of Virtual Game Simulation on Nursing Students' Knowledge and Skills Regarding Standard Infection Precautions
Brief Title: Virtual Game Simulation Effect on Nursing Students' Knowledge and Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Sakarya University (Other)
Responsible Party: Principal Investigator, Ebru Erek Kazan, Assoc.Prof., Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025/01
Record Dates: First submitted 2025-09-26; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Infection Control
Keywords: Infection Control; Standard infection precautions; Knowledge level; Nursing student; Skills; Virtual game simulation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Simulation Game (Experimental): The experimental group will be taught a theoretical course on standard infection precautions using the traditional method by the researcher. A knowledge test (pre-test) will be administered, practical training will be provided in the laboratory, and then a skills assessment (initial skill assessment) will be conducted. In addition to the traditional method, students in the experimental group will play a virtual game simulation through the Moodle Learning Management System. A knowledge (post-test) and skills assessment (post-skill assessment) will be conducted again one week later.
  Interventions: Other: Virtual Game Simulation Group and Conventional Education Group
- Traditional method (No Intervention): Students in the control group will be taught a theoretical lesson on standard infection precautions by the researcher using the traditional method. Following this, a knowledge test (pre-test) will be administered, followed by laboratory practice, and then a skills assessment (initial skill assessment). A week later, a knowledge (post-test) and skills assessment (post-skill assessment) will be administered again.

INTERVENTIONS:
Other: Virtual Game Simulation Group and Conventional Education Group — The intervention is an interactive virtual simulation game designed to teach standard precautions to nursing students. Unlike traditional skills lab training, the simulation presents realistic clinical scenarios in a digital environment, allowing students to repeatedly practice infection control procedures, receive immediate feedback, and utilize critical thinking skills in decision-making. This approach distinguishes the intervention from both traditional lectures and demonstration methods conducted during limited laboratory hours by providing experiential, student-centered, and technology-enhanced learning.
  Arms: Virtual Simulation Game

SUMMARY:
This study was designed as a randomized controlled experimental study to examine the effects of a virtual game simulation developed for standard infection precautions on the knowledge and skills of nursing students compared to a traditional education method. The study sample will consist of first-year nursing students studying in the Department of Nursing at Sakarya University, Faculty of Health Sciences in Turkey, during the Fall Semester of the 2025-2026 Academic Year. Written permissions for the conduct of the study obtained from the ethics committee and the institution. The study sample will consist of 130 students. The students will be randomly divided into two groups: 65 control and 65 experimental (virtual game simulation). Data will be collected using a "Descriptive Characteristics Form," "Knowledge Test on Standard Infection Precautions," "Skills Checklist for Medical Handwashing," "Skills Checklist for Donning and Doffing Sterile Gloves," "Skills Checklist for Donning and Doffing Personal Protective Equipment" and "Self-Debriefing Form." Knowledge and skills scores are expected to be higher in the experimental group, which received training supported by virtual game simulation in addition to traditional teaching methods, compared to the control group. The results of the study are expected to contribute to the literature.

DETAILED DESCRIPTION:
The study is a randomized controlled experimental study conducted to determine the effects of a virtual game simulation developed for standard infection precautions on the knowledge and skills of nursing students. The research will be conducted with first-year nursing students studying at the Department of Nursing, Faculty of Health Sciences, Sakarya University, in Turkey, during the Fall Semester of the 2025-2026 Academic Year. In order to conduct the research, written permission was obtained from the Sakarya University Social and Human Sciences Ethics Committee (Date:24.09.2025, Number:90/09) and the Sakarya University Faculty of Health Sciences, where the research will be conducted. In our study, with an effect size of 0.535 obtained from the source article, it was calculated that a total of 112 people, with a minimum of 56 people in each group, were required to study at 80% power and an α=0.05 error level. The G Power 3.1.9.7 package program was used in the sample calculation. In an experimental study, it is stated that keeping losses below 10% or 15% is important for reducing bias, and increasing the sample size is useful in controlling bias due to losses. Therefore, the number of students to be included in the sample was calculated as 130 (Experimental: 65, Control: 65) with a 15% probability of loss. Data in the study will be collected using the "Descriptive Characteristics Form," "Knowledge Test on Standard Infection Precautions," "Skill Checklists on Standard Infection Precautions," and "Self-Debriefing Form." A preliminary application will be conducted with second-year students at the university which the study will be conducted to evaluate the functionality of the data collection forms and the Moodle Learning Management System in the study. Necessary adjustments will be made to the forms and system operation based on the data obtained from the preliminary application. Randomization in determining the sample will be performed using the software program The R Project for Statistical Computing (Windows 2021, R version 4.1.2). Assignment to groups will be made in a way that ensures homogeneity based on gender and nursing department entrance scores.

Students will be divided into two groups: a virtual game simulation (experimental) and a control group, according to the order determined by the principal investigator. The researcher will made a theoretical lesson on standard infection precautions to students in the control group using a PowerPoint presentation using the methods of explanation, question-answer, and discussion. At the end of the lesson, the students will be administered a "Knowledge Test on Standard Infection Precautions" (pre-test) to measure their initial knowledge scores. The next day, students will be taken to the laboratory, where the researcher will demonstrate the skills of "Medical handwashing," "Sterile glove donning and doffing," and "Personal protective equipment donning and doffing" using a demonstration method, following the procedure steps. Subsequently, under the researcher's supervision, all students will be able to perform the specified skills. At the end of the laboratory lesson, students will be informed about the skill assessment to be performed the following day and will be provided with checklists containing the procedure steps for "Medical handwashing," "Sterile glove donning and doffing," and "Personal protective equipment donning and doffing." Students' skills will then be measured. To prevent bias, the researcher will not conduct a skill assessment; skill measurements will be conducted by two independent observers. Observers will not be informed of the students' group status. This will ensure that the observers are blinded to the study. The next day, in the laboratory, the students will be administered the "Skill Checklist for Medical Handwashing," the "Skill Checklist for Donning and Doffing Sterile Gloves," and the "Skill Checklist for Donning and Doffing Personal Protective Equipment" (initial skill assessment). No additional practice will be administered for seven days after the initial data from the control group students are collected. One week later, the students will be administered the "Standard Infection Precautions Knowledge Test" (posttest), and the skills "Medical Handwashing," "Sterile Glove Donning and Doffing," and "Personal Protective Equipment Donning and Doffing" (post-skill assessment) will be administered in the laboratory. After the control group data are collected, the experimental group will be assigned to the experimental group. This will prevent any interaction between the groups.

One week after the theoretical lesson was taught to the control group, the researcher will present a theoretical lesson on standard infection precautions using a PowerPoint presentation using the following methods: a brief explanation, question-answer, and discussion. At the end of the lesson, the students will be administered the "Knowledge Test on Standard Infection Precautions" (pre-test) to measure their initial knowledge scores. The next day, the students will be taken to the laboratory, where the researcher will demonstrate the skills of "Medical hand washing," "Sterile glove donning and doffing," and "Personal protective equipment donning and doffing" using a demonstration method, following the steps outlined. Then, under the researcher's supervision, all students will ensure that the specified skills are performed. At the end of the laboratory lesson, students will be informed about the skill assessment to be conducted the following day and will be provided with checklists containing the steps for "Medical hand washing," "Sterile glove donning and doffing," and "Personal protective equipment donning and doffing." The next day, in the laboratory, students' skills will be assessed by independent observers using the "Skills Checklist for Medical Handwashing," "Skills Checklist for Donning and Doffing Sterile Gloves," and "Skills Checklist for Donning and Doffing Personal Protective Equipment" (initial skill assessment). After the initial knowledge and skills assessment of the experimental group is completed, students in the experimental group will receive a 30-minute PowerPoint presentation in the classroom on how to log in to the Moodle Learning Management System and access the virtual game simulation. The researcher will email the students in the experimental group their username and password to access the virtual game simulation, which will be uploaded to the Moodle platform. Students will have access to the content of the virtual game simulation at their convenience and location for seven days. After all students complete the virtual game simulation, the researcher will ensure that all students in the experimental group complete the "Self-Debriefing Form" uploaded to Moodle. Students in the experimental group who experienced the virtual game simulation will be administered the "Standard Precautions Knowledge Test" (post-test) at the end of seven days, and their skills will be assessed in the laboratory using the "Medical Handwashing Skills Checklist," the "Sterile Glove Donning and Doffing Skills Checklist," and the "Personal Protective Equipment Donning and Doffing Skills Checklist" (post-skill assessment). After the experimental group's implementation is complete, students in the control group will also be able to play and benefit from the virtual game simulation.

ELIGIBILITY:
Inclusion Criteria:

* speak Turkish,
* are taking the Fundamentals of Nursing course for the first time,
* have no previous clinical experience,
* have internet access,
* have no visual, hearing, or motor skills limitations,
* owning a smartphone or computer will be included in the study.

Exclusion Criteria:

* Do not participate in virtual game simulations.

  * Do not attend the Fundamentals of Nursing course.
  * Do not attend the theoretical course on standard infection precautions.
  * Complete incomplete data collection forms,
  * Do not participate in any phase of the research; you will not be included in the study.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2025-10-07 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Knowledge | 1 month
  The study will use the "Knowledge Test on Standard Infection Precautions", developed by the researcher based on relevant literature, to measure students' knowledge of standard precautions. Knowledge Test on Standard Infection Precautions consists of a total of 30 questions, and a higher score indicates a higher level of knowledge. A minimum of 0 (zero) and a maximum of 30 points can be obtained on this knowledge test. In the control group, the test will be administered at the end of the conventional lesson (pre-test) and one week later (post-test). After collecting control group data, the experimental group will receive a theoretical lesson, followed by access to the virtual game simulation via Moodle for seven days. After completing the simulation, students will take the post-test. Knowledge scores will be compared between the virtual game simulation and control groups.
Skills | 3 months
  Nursing students' application of standard infection control precautions will be assessed before and after the intervention using a skills checklist developed by the researcher. The checklist will include practices such as medical handwashing, donning and doffing sterile gloves, and donning and doffing personal protective equipment. On the skill checklists, "2" points will be awarded for each correct step observed, "1" point for each incorrect/incomplete step, and "0 (zero)" points for each step not observed. Skill assessments will be conducted by two independent observers blinded to group allocation. The control group will receive a traditional theoretical lesson and laboratory practice on standard infection precautions, and end of the laboratory and one-week later skills assessments. The experimental group will receive the same training plus a seven-day virtual game simulation via Moodle, with skills reassessed end of the laboratory and one week later of virtual game simulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ordu Y, Caliskan N. The effects of virtual gaming simulation on nursing students' diagnosis, goal setting, and diagnosis prioritization: A randomized controlled trial. Nurse Educ Pract. 2023 Mar;68:103593. doi: 10.1016/j.nepr.2023.103593. Epub 2023 Mar 2. PMID 36871387
- [Background] Akın B, Kocoglu D. Randomized Controlled Trials. Journal of Hacettepe University Faculty of Nursing, 2017, 4(1):73-92.